CLINICAL TRIAL: NCT07049718
Title: Effect of Whole-body Vibration Training on Bone Mineral Density and Physical Performance in Patient With Renal Dialysis
Brief Title: Effect of Whole-body Vibration Training in Patients With Renal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Elsaid Ahmed Elsaid, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: whole body vibration training
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Renal Dialysis
Keywords: Renal Dialysis; Whole-Body Vibration; Bone Mineral Density; Physical Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration group (Experimental): Thirty male patients will receive whole body vibration twice / week for 12 weeks with duration from 30 to 60secound until reach 20 minutes and intensity begin from initially 5 HZ until reach 28 HZ gradually increase each 4 weeks in addition to medication (Red Blood Cell Stimulating Agents, Iron, Blood Pressure Medications, Phosphate Binders, Vitamins B and C, Calcitriol, Cinacalcet and Antibiotics).
  Interventions: Device: whole body vibration
- control group (No Intervention): Thirty male patients will receive their own medication only (Red Blood Cell Stimulating Agents, Iron, Blood Pressure Medications, Phosphate Binders, Vitamins B and C, Calcitriol, Cinacalcet and Antibiotics).

INTERVENTIONS:
Device: whole body vibration — Whole-body vibration (WBV) is a training method that uses mechanical vibration and external resistance loading to stimulate the body, causing muscle vibration and increasing central nervous system adaptations (Rittweger, 2010).
  Arms: whole body vibration group

SUMMARY:
To show the effect of whole-body vibration in physical performance in patients with renal dialysis.

DETAILED DESCRIPTION:
By now, safety and efficacy of WBV has not been investigated in patients with ESRD. Therefore, we performed this exploratory study in hemodialysis patients in order to elucidate potential effects of whole-body vibration exercise on physical performance and various biochemical markers in this condition. WBV is extensively studied as a means to prevent microgravity and immobility associated muscle wasting and bone loss in space flight and it is getting increasingly popular even among elderly.

Whole-body vibration exercise (WBVE) is a novel exercise protocol designed to prevent the loss of muscle strength and bone mineralization during the immobility and weightlessness of space flight.

A situation similar to HD. Vibration exercise uses high-frequency vibration of muscle groups causing positive feedback of the spinal reflex arc and resulting in high levels of muscle contraction to motor unit recruitment. There can be multiple physiological benefits from vibration exercise, including cardiovascular effects, bone health and muscle strength.

The advantages of WBV result from the combination of hardly any physical stress for the participants, short duration of intervention and a comparatively high effectiveness. means of exercise that can also be offered to those patients unable or unwilling to perform conventional training.

ELIGIBILITY:
Inclusion Criteria:

All patients that will be included in this study will meet the following criteria:

1. Body mass index (BMI) from 25.0 to 29.9 kg/m2.
2. Quitting smoking for more than 3 months.
3. Their age will be ranged from 60-70 years old.
4. Clinically and medically stable.
5. Hemodialysis treatment over at least 6 months before enrollment.
6. Patients with CKD (systolic blood pressure < 140 mmHg diastolic blood pressure < 90 mmHg and heart rate < 80 bpm).
7. The presence of kidney damage (i.e., albuminuria) or decreased kidney function (i.e. glomerular filtration rate (GFR) < 60 ml/min per 1-73 m2) for 3 months or more irrespective of clinical diagnosis.

   -

Exclusion Criteria:

Patients will be excluded if they have:

1. Patients with uncontrolled pulmonary disease.
2. Patients with vascular severe complication as critical limb ischemia.
3. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure.
4. Patients with severe musculoskeletal problems (e.g., severe knee osteoarthritis or post knee replacement surgeries).
5. Any patients who missed more than two weeks of the program or want to terminate the program.

   -

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
bone mineral density | 3 months
  Blood sample to take bone mineral density. (calcium & phosphorus)
physical performance | 3 months
  For participant's functional status will be evaluated by a series of physical performance tests

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Abdelmoniem, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Giza, Cairo University, Egypt

REFERENCES:
- [Background] Zierle-Ghosh A, Jan A. Physiology, Body Mass Index. 2023 Nov 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK535456/ PMID 30571077
- [Background] Zhanpeng F, Yan J, Fengrong Z, Sijie T. Estimation of peak oxygen pulse from body mass, resting heart rate, age, gender and systolic blood pressure in Chinese adults aged 20-39. Heliyon. 2023 Nov 4;9(11):e21912. doi: 10.1016/j.heliyon.2023.e21912. eCollection 2023 Nov. PMID 38027988
- [Background] Bai Y, Huang L, Yin X, Sun Q, Zhang F. Effects of whole-body vibration exercise on physical function in patients with chronic kidney disease: a systematic review and meta-analysis. BMC Nephrol. 2024 Jan 3;25(1):2. doi: 10.1186/s12882-023-03436-3. PMID 38172769
- [Background] van Heuvelen MJG, Rittweger J, Judex S, Sanudo B, Seixas A, Fuermaier ABM, Tucha O, Nyakas C, Marin PJ, Taiar R, Stark C, Schoenau E, Sa-Caputo DC, Bernardo-Filho M, van der Zee EA. Reporting Guidelines for Whole-Body Vibration Studies in Humans, Animals and Cell Cultures: A Consensus Statement from an International Group of Experts. Biology (Basel). 2021 Sep 27;10(10):965. doi: 10.3390/biology10100965. PMID 34681065
- [Background] Chen TK, Knicely DH, Grams ME. Chronic Kidney Disease Diagnosis and Management: A Review. JAMA. 2019 Oct 1;322(13):1294-1304. doi: 10.1001/jama.2019.14745. PMID 31573641
- [Background] Stenvinkel P, Carrero JJ, von Walden F, Ikizler TA, Nader GA. Muscle wasting in end-stage renal disease promulgates premature death: established, emerging and potential novel treatment strategies. Nephrol Dial Transplant. 2016 Jul;31(7):1070-7. doi: 10.1093/ndt/gfv122. Epub 2015 Apr 24. PMID 25910496
- [Background] Sietsema KE, Amato A, Adler SG, Brass EP. Exercise capacity as a predictor of survival among ambulatory patients with end-stage renal disease. Kidney Int. 2004 Feb;65(2):719-24. doi: 10.1111/j.1523-1755.2004.00411.x. PMID 14717947
- [Background] Seefried L, Genest F, Luksche N, Schneider M, Fazeli G, Brandl M, Bahner U, A Heidland A. Efficacy and safety of whole body vibration in maintenance hemodialysis patients - A pilot study. J Musculoskelet Neuronal Interact. 2017 Dec 1;17(4):268-274. PMID 29199185
- [Background] Howden EJ, Fassett RG, Isbel NM, Coombes JS. Exercise training in chronic kidney disease patients. Sports Med. 2012 Jun 1;42(6):473-88. doi: 10.2165/11630800-000000000-00000. PMID 22587820
- [Background] Rittweger J. Vibration as an exercise modality: how it may work, and what its potential might be. Eur J Appl Physiol. 2010 Mar;108(5):877-904. doi: 10.1007/s00421-009-1303-3. Epub 2009 Dec 12. PMID 20012646
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Marinho PEM, Rocha LG, Araujo Filho JC, Araujo AXP, Andrade MDA, Taiar R, Paiva DN, Dornelas de Andrade A. Effects of whole-body vibration on muscle strength, quadriceps muscle thickness and functional capacity in kidney transplant recipients: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:101-107. doi: 10.1016/j.jbmt.2020.10.005. Epub 2020 Oct 24. PMID 33992228
- [Background] Munhoz EC, Hollanda R, Vargas JP, Silveira CW, Lemos AL, Hollanda RM, Ribeiro JP. Flattening of oxygen pulse during exercise may detect extensive myocardial ischemia. Med Sci Sports Exerc. 2007 Aug;39(8):1221-6. doi: 10.1249/mss.0b013e3180601136. PMID 17762353
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Johnstone, L. M., Roshanravan, B., Rundell, S. D., Kestenbaum, B., Baker, S. F., Berry, D. L., & McGough, E. (2022). Instrumented and standard measures of physical performance in adults with chronic kidney disease. Journal of Acute Care Physical Therapy, 13(3), 110-118.
- [Background] James Myhre et al.,( 2023). "Stages of Kidney Disease and Treatment", https://www.verywellhealth.com/stages-of-kidney-disease-8303978..
- [Background] Isoyama N, Qureshi AR, Avesani CM, Lindholm B, Barany P, Heimburger O, Cederholm T, Stenvinkel P, Carrero JJ. Comparative associations of muscle mass and muscle strength with mortality in dialysis patients. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1720-8. doi: 10.2215/CJN.10261013. Epub 2014 Jul 29. PMID 25074839
- [Background] Housman, A. E., & Shropshire Lad, A. (2010). Incidence and prevalence. United States Renal Data System. 2010 Annual Data Report: atlas of chronic kidney disease and end-stage renal disease in the United States, 2.
- [Background] Beddhu S, Baird BC, Zitterkoph J, Neilson J, Greene T. Physical activity and mortality in chronic kidney disease (NHANES III). Clin J Am Soc Nephrol. 2009 Dec;4(12):1901-6. doi: 10.2215/CJN.01970309. Epub 2009 Oct 9. PMID 19820134
- [Background] Goodbred AJ, Langan RC. Chronic Kidney Disease: Prevention, Diagnosis, and Treatment. Am Fam Physician. 2023 Dec;108(6):554-561. PMID 38215416